CLINICAL TRIAL: NCT06884813
Title: Clinical Evaluation of a Single-Shade, Color-Adjusting Composite Resin Following In-Office Dental Bleaching: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Color-Adjusting Composite Resin Following In-Office Dental Bleaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250033
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Composite Resins
Keywords: Single-shade composite; Bleaching; clinical trial; Shade matching
MeSH Terms: interventions — Hydrogen Peroxide; Erythrocyte Count

STUDY DESIGN:
Intervention Model Description: Split mouth study design, patients will be assigned to two different treatment protocols.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) The patients who participated in the study and the assessor of the treatment outcome do not know the type of treatment procedure received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Conventional RBC) (Experimental): In office bleaching for teeth restored using conventional multishade nanohybrid resin based composite (RBC).
  Interventions: Drug: Conventional nanohybrid multishade composite and hydrogen peroxide 40% in-Office Tooth Whitening System
- Test group (RBC with CAP) (Experimental): In office bleaching for teeth restored using Omnichroma (single shade) composite with color adjustment postential (CAP).
  Interventions: Drug: Single shade nanohybrid composite and hydrogen peroxide 40% in-Office Tooth Whitening System

INTERVENTIONS:
Drug: Conventional nanohybrid multishade composite and hydrogen peroxide 40% in-Office Tooth Whitening System — Teeth restored with conventional multi shade nanohybrid Resin Based Composite (RBC) Filtek Z350Xt (3M ESPE, San Paul, MN, USA) subjected to bleaching using Opalescence Boost 40% In-Office Tooth Whitening System (Ultradent, Utah, USA)
  Other Names: Conventional resin based composite (RBC) and Hydrogen perioxide 40%
  Arms: Control group (Conventional RBC)
Drug: Single shade nanohybrid composite and hydrogen peroxide 40% in-Office Tooth Whitening System — Teeth restored with One-shade Resin Based Composite (Omnichroma, Tokuyama Dental, Tokio, Japan) subjected to bleaching using Opalescence Boost 40% In-Office Tooth Whitening System (Ultradent, Utah, USA)
  Other Names: RBC with color adjustment potential (CAP) and Hydrogen perioxide 40%
  Arms: Test group (RBC with CAP)

SUMMARY:
One challenge faced by dental professionals is that, unlike natural tooth structure, composite restorations do not lighten when exposed to bleaching agents. As a result, functional restorations may need replacement after bleaching to match the newly whitened teeth. However, replacing a composite restoration can lead to unnecessary removal of tooth structure, potentially weakening the tooth and increasing its susceptibility to further iatrogenic damage. This study will investigate the ability of Omnichroma restorations to shade-match tooth structure after bleaching.

The null hypotheses will be:

1. Single-shade RBC will not exhibit similar shade and optical behavior to conventional RBC across all anterior restorations following bleaching.
2. Patient satisfaction regarding color blending between the restoration and tooth structure will not differ according to the type of material used.
3. Dentist satisfaction regarding color blending between the restoration and tooth structure will not differ according to the type of material used.

DETAILED DESCRIPTION:
Selecting the proper shade for a restoration is of vital importance for achieving optimal aesthetic results. However, shade selection can be time-consuming, somewhat subjective, and heavily reliant on the clinician's visual judgement.

This study will explore the ability of Omnichroma restorations to shade match tooth structure after bleaching. Patients visiting the JUST dental clinics who have at least two anterior restorations (one Omnichroma restoration and one multi-shade nanohybrid composite restoration) will be recruited for this study. The calculated sample size for the study is 240 teeth.

The shade and the L*a*b* scores will be recorded using spectrophotometer prior to bleaching and after bleaching. Two blinded, calibrated dentists will independently evaluate the resulting shade outcomes and assess the degree of color match between the restorations and the adjacent teeth after bleaching. This assessment will be categorized as either match or no match. The patient's satisfaction will also be recorded two weeks after bleaching.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to come back for follow-up appointments.
2. Patients who are willing to sign an informed consent form.
3. Patients with well documented clinical records and have at least two anterior restorations (both Omnichroma and conventional multi-shade nanohybrid composite.)
4. Patients aged 18 years or older.
5. Patients with good oral hygiene
6. Patients with vital teeth.
7. Patients who are willing to have the restorations replaced later if necessary if there is a color mismatch after bleaching treatment.

Exclusion Criteria:

1. Individuals with severe bruxism or periodontal disease.
2. Patients with non-vital teeth restored with composite fillings.
3. Patients with severe tooth discoloration.
4. Patients with fluorosis or tetracycline staining.
5. Heavy smokers.
6. Pregnant or nursing women.
7. Patients undergoing orthodontic treatment.
8. Patients with enamel or dentin deformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Color measurements using digital spectrophotometer VITA Easyshade V. | One year
  The colour measurements will be taken at first session for each tooth in specific points as follow:
  One reading from middle part of tooth Three readings at three points around the restoration and 1 mm away from its margins.
  To give a chance for tooth rehydration and final color optimization, a new reading will be obtained from the middle portion of the restoration after one week.
  The color difference (∆E00) between the tooth structure around the restoration and the restoration itself will be calculated.
  The color difference (∆E00) between the tooth and restoration will be compared between the control and test groups.
  The final ΔE00 value itself has no physical unit. It is just a numerical representation of color difference.
Subjective or Patient satisfaction | One year
  Patient satisfaction regarding color blending between the restoration and tooth surface will be recorded after one week using visual analogue scale (VAS).
  The scale is a horizontal line with 10 digits, where 0 (on the right) represents total dissatisfaction with color blending between the tooth and restoration, and 10 (on the left) indicates complete satisfaction.
  Patients will mark their satisfaction with the color matching and blending of the restoration on the VAS.
  Measurements will be categorized as follows:
  Poor: VAS values from 0 to 5 Good: VAS values from 5.1 to 10
Objective or dentists satisfaction | One year
  Photographs of the restored teeth will be taken under a standardized setup using a Canon 250D DSLR camera, a Sigma 105 mm macro lens, and a Meike MK-14EXT TTL macro ring flash.
  The images will be evaluated by two calibrated dentists who are blinded to the restoration material. Blending with the tooth surface will be assessed using VAS, with the assessors marking their evaluation on the scale.
  Measurements will be divided according following criteria:
  Poor: VAS values ranging from 0-5. Good :VAS values ranging from 5.1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villarroel M, Fahl N, De Sousa AM, De Oliveira OB Jr. Direct esthetic restorations based on translucency and opacity of composite resins. J Esthet Restor Dent. 2011 Apr;23(2):73-87. doi: 10.1111/j.1708-8240.2010.00392.x. Epub 2011 Feb 25. PMID 21477031
- [Background] Hafez R, Ahmed D, Yousry M, El-Badrawy W, El-Mowafy O. Effect of in-office bleaching on color and surface roughness of composite restoratives. Eur J Dent. 2010 Apr;4(2):118-27. PMID 20396441
- [Background] Forabosco E, Consolo U, Mazzitelli C, Kaleci S, Generali L, Checchi V. Effect of bleaching on the color match of single-shade resin composites. J Oral Sci. 2023 Oct 1;65(4):232-236. doi: 10.2334/josnusd.23-0159. Epub 2023 Aug 3. PMID 37532526
- [Background] AlHabdan A, AlShamrani A, AlHumaidan R, AlFehaid A, Eisa S. Color Matching of Universal Shade Resin-Based Composite with Natural Teeth and Its Stability before and after In-Office Bleaching. Int J Biomater. 2022 Oct 26;2022:8420890. doi: 10.1155/2022/8420890. eCollection 2022. PMID 36341131